CLINICAL TRIAL: NCT02049996
Title: Is There a Difference in Pain and Quality of Life Following Vaginal Hysterectomy With Vaginal Reconstruction Compared to Robotic Colpopexy? A Prospective Cohort Study
Brief Title: Difference in Pain, Quality of Life Following Vaginal Hysterectomy With Vaginal Reconstruction Versus Robotic Colpopexy?
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 13090-13-060
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Pelvic Organ Prolapse
Keywords: Quality of life; Robotic surgery; Vaginal surgery; Prolapse repair; Vaginal hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Robotic-assisted prolapse repair: Subjects already scheduled for robotic-assisted prolapse repair in conjunction with vaginal hysterectomy
- Vaginal prolapse repair: Subjects already scheduled for vaginal prolapse repair in conjunction with vaginal hysterectomy.

SUMMARY:
The purpose of this study is to to determine if there is a difference in patient related outcomes of pain and quality of life following vaginal hysterectomy with vaginal prolapse repair compared to robotic-assisted repair.

We hypothesize that pain and quality of life following robotic-assisted repair will be similar to that following vaginal reconstruction, when performed in conjunction with vaginal hysterectomy.

DETAILED DESCRIPTION:
Since the introduction of the DaVinci robotic system (Intuitive Surgical, Sunnyvale, CA), there has been considerable debate regarding its use, cost-effectiveness, and subsequent impact on patient care. While some studies have examined surgical outcomes and analyzed costs of this technique compared to open, laparoscopic, and vaginal approaches, it remains unclear whether one route is superior.

Indeed, data evaluating robotic-assisted and laparoscopic approaches to hysterectomy have shown similar patient results, but some reports note higher costs and longer operating times with robotics. Others suggest contrary information, with comparable surgical time, reduced blood loss, shorter hospital stay, and lower rate of conversion to laparotomy using robotic-assisted hysterectomy compared to laparoscopic or abdominal. Research contrasting robot-assisted laparoscopic myomectomy with abdominal myomectomy posit greater cost associated with the robotic procedure, but enhanced benefit of decreased blood loss, complication rates, and length of stay.

However, these issues have not been explored in urogynecologic patients. A single study comparing robotic versus vaginal urogynecologic procedures in elderly women showed robotic surgery to be associated with fewer postoperative complications than the vaginal route. Nevertheless the procedures were not always performed in conjunction with hysterectomy, and the analysis was retrospective.

In our practice, vaginal hysterectomy is the preferred method when correcting uterovaginal prolapse. We then address the reconstruction either vaginally or robotically. Vaginal repairs are comprised of the following: a vaginal vault suspension using the uterosacral ligaments, enterocele repair, anterior repair, and posterior/rectocele repair. The robotic procedure performed is a robotic sacral colpopexy using lightweight, polypropylene mesh, as well as a posterior/rectocele repair transvaginally. Both of these techniques are well-researched, effective approaches to addressing prolapse in a durable way. However, it is not clear whether one is superior in patient-related quality of life outcomes. We seek to compare patient quality of life by assessing differences in subjective impressions of pain following these procedures

ELIGIBILITY:
Inclusion Criteria:

* patients of Cincinnati Urogynecology Associates
* aged 18-90
* planning to undergo a vaginal hysterectomy with robotic or vaginal reconstructive surgery for pelvic organ prolapse as well as a posterior/rectocele repair, with or without a suburethral sling or ovarian removal.
* undergoing general anesthesia
* able to speak and read English
* able to understand the informed consent statement

Exclusion Criteria:

* scheduled for repairs not involving a hysterectomy
* use of mesh in the vaginal prolapse repair
* obliterative procedures to the vagina
* concurrent removal of a suburethral sling
* anterior, posterior or apical vaginal mesh kit at the time of their surgery
* performance of vaginal 'relaxing incisions' at the time of vaginal surgery
* concurrent anal incontinence repair such as a sphincteroplasty
* presence of uterine, cervical or ovarian malignancy
* use of regional anesthesia for their surgery.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have been scheduled for a vaginal hysterectomy with either vaginal or robot-assisted prolapse repairs with Cincinnati Urogynecology Associates will be approached for participation in the study.
  Eligible subjects are patients of Cincinnati Urogynecology Associates, aged 18-90, planning to undergo a vaginal hysterectomy with robotic or vaginal reconstructive surgery for pelvic organ prolapse, as well as a posterior/rectocele repair, with or without a suburethral sling or ovarian removal. All subjects will undergo general anesthesia. Eligible subjects must be able to speak and read English, and be able to understand the informed consent statement.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of pain on the morning of post-operative day 1 | One day (the day after surgery)
  Subjective assessment of pain on the morning of post-operative day 1, prior to discharge, on a 150 mm visual analog scale (Surgical Pain Scale) The average pain that day at rest and the WORST pain that day will be the primary outcomes of pain.

SECONDARY OUTCOMES:
Subjective assessment of pain at 2 week postoperative visit and 6 week postoperative visit | 2 week postoperative visit
  Subjective assessment of pain at 2 week postoperative visit and 6 week postoperative visit on a 150 mm visual analog scale (Surgical Pain Scale).
Subjective assessment of pain at 2 week postoperative visit and 6 week postoperative visit | 6 week postoperative visit
  Subjective assessment of pain at 2 week postoperative visit and 6 week postoperative visit on a 150 mm visual analog scale (Surgical Pain Scale).
Quality of life at baseline, 2 week postoperative, and 6 week postoperative visit | 1 day (Baseline, day of surgery)
  General Health Survey- Short Form 12 looking at quality of life at baseline, 2 week postoperative, and 6 week postoperative visit.
Quality of life at baseline, 2 week postoperative, and 6 week postoperative visit. | 2 week postoperative visit
  General Health Survey- Short Form 12 looking at quality of life at baseline, 2 week postoperative, and 6 week postoperative visit.
Quality of life at baseline, 2 week postoperative, and 6 week postoperative visit. | 6 week postoperative visit
  General Health Survey- Short Form 12 looking at quality of life at baseline, 2 week postoperative, and 6 week postoperative visit.
Intraoperative time | Intraoperative
  Length of surgery
Estimated blood loss | Intraoperative
  Estimated blood loss during surgery.
Surgical complications | Intraoperative
  Complications that occur during surgery.
Voiding trial results | 1 day (day after surgery)
  Results of voiding trial which assesses postoperative bladder function.
Hospital length of stay | 1-2 days
  Length of stay in the hospital for surgery and postoperative care.
POP-Q preoperatively and postoperatively | several weeks
  Comparison measurement of prolapse using pelvic organ prolapse quantification scale (POP-Q) preoperatively and postoperatively.
Hemoglobin/hematocrit measurement | 1 day (postoperative day 1)
  Measurement of blood count (hemoglobin/hematocrit levels) on postoperative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren B. Westermann, DO, Principal Investigator — TriHealth Good Samaritan Hospital
Locations (1):
- TriHealth Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payne TN, Dauterive FR. A comparison of total laparoscopic hysterectomy to robotically assisted hysterectomy: surgical outcomes in a community practice. J Minim Invasive Gynecol. 2008 May-Jun;15(3):286-91. doi: 10.1016/j.jmig.2008.01.008. Epub 2008 Mar 6. PMID 18439499
- [Background] Shashoua AR, Gill D, Locher SR. Robotic-assisted total laparoscopic hysterectomy versus conventional total laparoscopic hysterectomy. JSLS. 2009 Jul-Sep;13(3):364-9. PMID 19793478
- [Background] Orady M, Hrynewych A, Nawfal AK, Wegienka G. Comparison of robotic-assisted hysterectomy to other minimally invasive approaches. JSLS. 2012 Oct-Dec;16(4):542-8. doi: 10.4293/108680812X13462882736899. PMID 23484561
- [Background] Advincula AP, Xu X, Goudeau S 4th, Ransom SB. Robot-assisted laparoscopic myomectomy versus abdominal myomectomy: a comparison of short-term surgical outcomes and immediate costs. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):698-705. doi: 10.1016/j.jmig.2007.06.008. PMID 17980329
- [Background] Bump RC, Mattiasson A, Bo K, Brubaker LP, DeLancey JO, Klarskov P, Shull BL, Smith AR. The standardization of terminology of female pelvic organ prolapse and pelvic floor dysfunction. Am J Obstet Gynecol. 1996 Jul;175(1):10-7. doi: 10.1016/s0002-9378(96)70243-0. PMID 8694033
- [Background] McCarthy M Jr, Chang CH, Pickard AS, Giobbie-Hurder A, Price DD, Jonasson O, Gibbs J, Fitzgibbons R, Neumayer L. Visual analog scales for assessing surgical pain. J Am Coll Surg. 2005 Aug;201(2):245-52. doi: 10.1016/j.jamcollsurg.2005.03.034. PMID 16038823
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135
- [Result] Sarlos D, Kots L, Stevanovic N, Schaer G. Robotic hysterectomy versus conventional laparoscopic hysterectomy: outcome and cost analyses of a matched case-control study. Eur J Obstet Gynecol Reprod Biol. 2010 May;150(1):92-6. doi: 10.1016/j.ejogrb.2010.02.012. Epub 2010 Mar 5. PMID 20207063
- [Result] Saceanu S, Cela V, Surlin V, Angelescu CM, Patrascu S, Georgescu I, Genazzani A. Hysterectomy for benign uterine pathology: comparison between robotic assisted laparoscopy, classic laparoscopy and laparotomy. Chirurgia (Bucur). 2013 May-Jun;108(3):346-50. PMID 23790783
- [Result] Patzkowsky KE, As-Sanie S, Smorgick N, Song AH, Advincula AP. Perioperative outcomes of robotic versus laparoscopic hysterectomy for benign disease. JSLS. 2013 Jan-Mar;17(1):100-6. doi: 10.4293/108680812X13517013317914. PMID 23743379
- [Result] Robinson BL, Parnell BA, Sandbulte JT, Geller EJ, Connolly A, Matthews CA. Robotic versus vaginal urogynecologic surgery: a retrospective cohort study of perioperative complications in elderly women. Female Pelvic Med Reconstr Surg. 2013 Jul-Aug;19(4):230-7. doi: 10.1097/SPV.0b013e318299a66c. PMID 23797528
- [Result] Crisp CC, Bandi S, Kleeman SD, Oakley SH, Vaccaro CM, Estanol MV, Fellner AN, Pauls RN. Patient-controlled versus scheduled, nurse-administered analgesia following vaginal reconstructive surgery: a randomized trial. Am J Obstet Gynecol. 2012 Nov;207(5):433.e1-6. doi: 10.1016/j.ajog.2012.06.040. Epub 2012 Jun 20. PMID 22863282
- [Derived] Westermann LB, Crisp CC, Mazloomdoost D, Kleeman SD, Pauls RN. Comparative Perioperative Pain and Recovery in Women Undergoing Vaginal Reconstruction Versus Robotic Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):95-100. doi: 10.1097/SPV.0000000000000368. PMID 28067743